CLINICAL TRIAL: NCT00181896
Title: Open-Label Study of Bupropion SR for Major Depression and Depression NOS in Children and Adolescents With Bipolar and Bipolar Spectrum Disorder
Brief Title: Bupropion SR for Major Depression and Depression NOS in Children and Adolescents With Bipolar Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated due to lack of recruitment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Joseph Biederman, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-P-001727
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Depression; Bipolar Disorder
Keywords: depression; bipolar disorder; children; bupropion SR
MeSH Terms: conditions — Depression; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bupropion SR — Open-label prescription of Bupropion SR for 8 weeks.

SUMMARY:
This is an 8-week open label study of bupropion SR in the treatment of youth with bipolar depression with adequate mood stabilization. All youth will be closely monitored for treatment emergent manic activation and drug-drug interactions with ongoing antimanic agents.

The main objective of this study is to assess the safety and effectiveness of bupropion SR in the treatment of bipolar depression in children and adolescents.

DETAILED DESCRIPTION:
While anti-manic agents can effectively control manic symptoms, bipolar patients frequently continue to struggle with residual depressive symptomatology that can be associated with severe morbidity and suicidality. Because antidepressants can activate manic symptoms in bipolar patients with depression, the treatment of bipolar depression poses unique and challenging therapeutic dilemmas Thus, the identification of appropriate safe and effective treatment strategies for the management of depression in bipolar youth is particularly taxing considering that pediatric mania is predominantly mixed with a strong depressive component. A recent study in our program of bupropion SR in 30 adults with ADHD and Bipolar disorder, treatment with bupropion SR was extremely well tolerated and was not associated with activation of manic symptoms. Because bupropion has not been evaluated in the treatment of bipolar depression in youth, there is a pressing need to evaluate its effectiveness and safety in the context of a treatment protocol aimed at carefully evaluating this issue.

This is an 8-week open label study of bupropion SR in the treatment of youth with bipolar depression with adequate mood stabilization. All youth will be closely monitored for treatment emergent manic activation and drug-drug interactions with ongoing antimanic agents.

The main objective of this study is to assess the safety and effectiveness of bupropion SR in the treatment of bipolar depression in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 6 to 17 with a diagnosis of current depression with bipolar disorder based on clinical assessment and confirmed by structured diagnostic interview plus an initial Hamilton rating scale score >17 and a Young Mania Rating Score of < 15.
* Children will only be allowed to participate in the trial if they have had mood stabilization on a steady dose of medication for at least 2 months. By mood stabilization we mean as determined by principle investigator, evaluator clinician, and as confirmed by KSADS.
* Subject and parent must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
* Subjects and their legal representative must be considered reliable.
* Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative must sign an informed consent document and the subject must sign an informed assent document.
* Subject must be able to participate in mandatory blood draws.
* Subject must be able to swallow pills.

Exclusion Criteria:

Subjects with chronic medical illness, DSM-IV substance dependence within the past month, pregnant or nursing female subjects will be excluded from this study.

* Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
* Serious, unstable illness including hepatic, renal, gastroenterological, respiratory, cardiovascular, endocrine, neurologic, immunologic, or hematologic disease.
* History of severe allergies or multiple adverse drug reactions.
* Non-febrile seizures without a clear and resolved etiology.
* Leukopenia or history of leukopenia without a clear and resolved etiology.
* Judged clinically to be at serious suicidal risk.
* Acute Psychosis
* Any other concomitant medication with primarily central nervous system activity other than specified in Concomitant Medication portion of the protocol.
* History of intolerance or non-response to bupropion.
* Treatment with nonreversible monoamine oxidase inhibitor within 2 weeks prior to initiation of study.
* Current diagnosis of schizophrenia.
* History of head trauma
* CNS tumor
* Diabetic treated with oral hypoglycemics or insulin
* Current or prior diagnosis of bulimia or anorexia

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2005-01; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
reduction in depression symptoms assessed by | baseline to 8 weeks
Children's Depression Rating Scale | baseline to 8 weeks
Hamilton Depression Rating scale (HAM-D) | baseline to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States